CLINICAL TRIAL: NCT06653777
Title: Phase II Trial Evaluating the Efficacy of Pemigatinib in Patients With Recurrent and/or Metastatic Solid Tumor Harboring a FGFR Alteration
Brief Title: Efficacy of Pemigatinib in Patients With Solid Tumors Characterized by an Alteration of the Gene FGFR in Tumor Cells
Acronym: AcSé PEMI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: National Cancer Institute, France (Other Government); Incyte BioSciences France (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC-GMP-2305; 2024-512729-10-00 (EU CTIS Number)
Record Dates: First submitted 2024-10-21; First posted 2024-10-22 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Solid Tumor, Miscellaneous
Keywords: pemigatinib; FGFR alteration
MeSH Terms: interventions — pemigatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pemigatinib (Experimental): Pemigatinib will be administered orally once daily for 2 weeks followed by a 1-week off (intermittent schedule 2/1).
  Interventions: Drug: Pemigatinib

INTERVENTIONS:
Drug: Pemigatinib — Pemigatinib will be administered orally once daily for 2 weeks followed by a 1-week off (intermittent schedule 2/1).
  Other Names: Pemazyre®

SUMMARY:
Alterations in the fibroblast growth factor receptor (FGFR) gene are involved in the development of cancer. These anomalies are found at very variable frequencies (from less than 1% to around 10%) in cancers of the bile ducts, bladder, uterus, brain, ovary, lung, airways, digestive tract, breast, etc.

Pemigatinib is an anti-cancer drug that acts on cells with alterations in the FGFR gene. It is used in Europe to treat people with biliary tract cancer who carry a specific FGFR alteration.

However, in various clinical trials, pemigatinib has shown interesting activity in a number of patients with different cancers presenting with an alteration in the FGFR gene. This treatment could therefore be effective in several types of cancer where an alteration in the FGFR gene is detected.

The aim of this clinical trial is to learn if pemigatinib works to treat patients with recurrent and/or metastatic cancer (whatever the type of cancer excluding blood cancers and those already treated with pemigatinib) presenting an alteration in the FGFR gene.

Patients will:

* Take oral pemigatinig in 3-week cycles (every day for 2 weeks followed by one week without pemigatinib) as long as they benefit from it.
* Visit the clinic once every 3 weeks for checkups and tests during the treatment period
* Visit the clinic once every 3 months for checkups after stopping treatment for at least 12 months.

DETAILED DESCRIPTION:
Anti-cancer treatments targeting abnormalities in the FGFR gene are currently marketed for biliary tract and bladder cancers, having demonstrated a certain degree of efficacy. In clinical trials, these drugs have shown promising signs of efficacy in other types of cancer with the same FGFR gene alterations.

All the patients included in this clinical trial will receive pemigatinib. The expected benefit for patient is the control of the disease through stabilization, reduction or even disappearance of the cancer and related symptoms.

The risks are mainly related to the adverse effects of the drug. The regular monitoring offered by the hospital and the additional examinations (such as more regular X-ray examinations, eye tests and blood tests) may constitute constraints. However, this monitoring and these examinations are carried out in order to better monitor and treat the effects of pemigatinib for both patient safety and the course of the disease.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed solid tumor
2. Patient with locally recurrent unresectable and/or advanced or metastatic disease harbouring a FGFR1,2,3 fusion/rearrangement or mutation
3. Age ≥ 18 years
4. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
5. Patient for whom there is no appropriate therapeutic alternative and for whom a FGFR inhibitor is indicated by the institution or the regional multidisciplinary consultation meeting and who may derive a benefit, according to the physician assessment
6. Estimated life expectancy >3 months
7. Measurable disease according to response evaluation criteria in solid tumours version 1.1 (RECIST1.1), whatever the disease location. Tumor lesions located in a previously irradiated area, or in an area subjected to other loco-regional therapy, are considered measureable if progression has been clearly demonstrated in the lesion.
8. Availability of 2 pre-treatment tumor evaluations performed with an interval of at least 4 weeks and no more than 3 months between the examinations (CT or MRI, but same technics for both) and without any cancer treatment during this period
9. Patient with a minimal trend at 0.1 mm/day increase in tumor growth kinetics between pre-treatment and baseline scan, as assessed by the investigator
10. Adequate hematologic function: Absolute neutrophil count (ANC) > 1.5 x 10⁹ /L; platelets > 75 x 10⁹ /L; haemoglobin > 9.0 g/dL. Transfusion is allowed with a 2-week washout period before treatment initiation
11. Adequate hepatic function: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2,5 x upper limit of normal (ULN) (≤ 5 x ULN for liver metastasis); total bilirubin < 1.5 x ULN (< 2.5 x ULN if Gilbert's syndrome or liver metastasis); alkaline phosphatase (ALP) < 3 x ULN
12. Adequate renal function: serum creatinine clearance > 30 mL/minute based on Cockcroft-Gault formula
13. Value of serum phosphate ≤ ULN and value of serum calcium within institutional normal range (or serum albumin-corrected calcium within normal range when serum albumin is outside of the normal range)
14. Potassium levels within institutional normal range; supplementation can be used to correct potassium level during the screening.
15. Men, and women of childbearing potential must agree to use adequate contraception for the duration of trial participation and for at least one week after the last dose of pemigatinib. Men must also agree to not donate sperm and women must agree to not donate oocytes during the specified period
16. Women of childbearing potential must have a negative serum pregnancy test performed within 14 days before treatment initiation
17. Patient is affiliated to a social security system
18. Patient must have signed a written informed consent form prior to any trial specific procedures. When the patient is physically unable to give their written consent, a trusted person of their choice, independent from the investigator or the sponsor, can confirm in signing the patient's consent

Exclusion Criteria:

1. Hematologic malignancies
2. Known hypersensitivity or severe reaction to pemigatinib or excipients of pemigatinib
3. Patient with a disease and a FGFR alteration covered by a marketed indication for any selective FGFR inhibitor (e.g cholangiocarcinoma with FGFR2-fusion or a FGFR mutation are not eligible, while FGFR1 or 3 fusion are eligible)
4. Patient who received prior selective FGFR inhibitor
5. Patient who can be included in a recruiting study assessing FGFR inhibitor (including pemigatinib)
6. Current evidence of clinically significant corneal or retinal disorder as confirmed by ophthalmologic examination
7. Other current malignancy, with the exception of adequately treated cone-biopsied in situ carcinoma of the cervix uteri and basal or squamous cell carcinoma of the skin. Cancer survivors, who have undergone potentially curative therapy for a prior malignancy, have no evidence of that disease for 5 years or more and are deemed at negligible risk for recurrence, are eligible for the trial
8. History of calcium and phosphate hemostasis disorder or systemic mineral imbalance with ectopic calcification of soft tissues (exception: commonly observed calcifications in soft tissues such as skin, kidney tendon, or vessels due to injury, disease, or aging in the absence of systemic mineral imbalance)
9. Significant gastrointestinal disorder(s) that could interfere with absorption, metabolism, or excretion of pemigatinib
10. Inability to swallow and retain oral medication
11. Clinically significant or uncontrolled cardiac disease, including unstable angina, acute myocardial infarction within 6 months from Day 1 of study drug/treatment administration, New York Heart Association Class III or IV congestive heart failure, and uncontrolled arrhythmia (participants with pacemaker or with atrial fibrillation and well-controlled heart rate are allowed)
12. History or presence of an abnormal electrocardiogram that, in the investigator's opinion, is clinically meaningful. A screening QTcF interval > 480 ms is excluded.
13. Evidence of active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection (defined as elevated transaminases or cirrhosis); chronic HBV/HCV infection with no cirrhosis and no elevated transaminases is allowed
14. Known HIV infection except if undetectable viral load
15. Other active chronic or current infectious disease requiring systemic antibiotic, antifungal, or antiviral treatment within 2 weeks before enrollment (participants with asymptomatic chronic infections on prophylactic treatment are allowed)
16. Prior anticancer therapy, including radiotherapy, endocrine therapy, immunotherapy, chemotherapy or other investigational agents within the last 4 weeks (6 weeks for nitrosoureas and mitomycin C). A 1-week washout is permitted for palliative radiation to non-central nervous system disease. Patients must have recovered (≤ Grade 1) from AEs from previously administered therapies or local treatments before treatment initiation (excluding alopecia, anemia and decreased creatinine clearance)
17. Use of any potent CYP3A4 inhibitors or inducers or moderate CYP3A4 inducers within 14 days or five half-lives (whichever is shorter) before the first dose of study drug
18. Any condition which in the Investigator's opinion makes it undesirable for the subject to participate in the trial or which would jeopardize compliance with the protocol
19. Inability or unlikeliness of the participant to comply with the dose schedule or with the medical evaluations and follow-up required by the trial because of geographic, familial, social, or psychological reasons
20. Women who are pregnant or breastfeeding
21. History of hypovitaminosis D requiring supraphysiologic doses (eg, 50,000 international unit (IU)/weekly) to replenish the deficiency.
22. Participation in another therapeutic trial within the 30 days prior to inclusion
23. Individuals deprived of liberty or placed under protective custody or guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-27 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Tumor regression | From enrollment to disease progression, up to 42 months
  Proportion of patients experiencing an objective response or at least a 30% decrease in tumor growth kinetics at disease progression on study treatment as compared to the one calculated from the two pre-treatment tumor evaluations. The tumor kinetics variation is measured by the tumor growth ratio defined as the ratio of the slope of tumor growth on treatment (between the nadir and disease progression) and the slope of tumor growth before treatment. The sum of the diameters of target lesions according to RECIST 1.1 will be calculated on each patient's imaging by the Blinded Independent Central Review (BICR).

SECONDARY OUTCOMES:
Overall response rate (ORR) | From enrollment to the progression, up to 42 months
  ORR is defined as the proportion of patients with a complete response (CR) or a partial response (PR) as best overall response during the study, based on RECIST1.1, as assessed by the BICR and by the physician.
Clinical benefit rate (CBR) | From enrollment to the progression, up to 42 months
  CBR defined as the proportion of patients with a CR, a PR, or a stable disease (SD) lasting ≥ 24 weeks (6 months) as best overall response during the study, based on RECIST1.1, as assessed by the BICR and by the physician.
Duration of response (DoR) | From enrollment to the progression, up to 42 months
  Duration of response (DoR) measured in responder patients from the time of first documented response (CR or PR) until the first documented disease progression (according to RECIST1.1) or death due to any cause, as assessed by the BICR and by the physician.
Progression-free survival (PFS) | From enrollment to disease progression or death, up to 42 months
  PFS measured from the date of inclusion to the date of event defined as the first documented disease progression (according to RECIST1.1) or death from any cause, whichever occurs first as assessed by the BICR and by physicians. Patients with no event at the time of analysis will be censored at the date of last adequate tumor assessment.
Time to treatment failure (TTF) | From enrollment to the end of treatment (or up to 42 months)
  TTF defined as the time from the date of inclusion to the date of permanent study treatment discontinuation (any cause, including disease progression, treatment toxicity and death, withdrawal of consent). Patients without treatment failure at the time of the analysis will be censored at the date of last tumor assessment.
Overall survival (OS) | From enrollment to death (or up to 42 months)
  OS measured from the date of inclusion to the date of death from any cause. Patients who are alive at the time of analysis (including lost to follow-up) will be censored at the date of last contact.
Safety and tolerability of pemigatinib | From enrollment to the end of treatment (up to 42 months)
  Safety and tolerability, as assessed by the occurrence of treatment-emergent and treatment-related adverse events according to the National Cancer Institute-Common Terminology Criteria for Adverse Events version 5 (NCI-CTCAE v5). The NCI-CTCAE v5 is widely accepted in the community of oncology research as the leading rating scale for adverse events. This scale, divided into 5 grades (1 = "mild", 2 = "moderate", 3 = "severe", 4 = "life-threatening", and 5 = "death") determined by the investigator, will make it possible to assess the severity of the disorders.
Quality of life questionnaire - Core 30 (QLQ-C30) | At baseline, at 3 and 6 months during treatment and at the end of treatment
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials.
  The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe LE TOURNEAU, Pr, Principal Investigator — Institut Curie Paris
Locations (6):
- France (6):
  - CHU de BREST, Brest
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - CHU Poitiers, Poitiers
  - CHU Saint Etienne, Saint-Priest-en-Jarez
  - Institut de Cancerologie de Lorraine, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients.